CLINICAL TRIAL: NCT03650218
Title: A Prospective, Open Label, Dose-escalating, Multicenter Clinical Investigation to Evaluate the Safety and Effectiveness of THIODERM STRONG in the Correction of Nasolabial Folds.
Brief Title: Safety and Effectiveness of THIODERM STRONG in the Correction of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPH-201-201334
Record Dates: First submitted 2018-08-09; First posted 2018-08-28 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Correction of Nasolabial Folds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THIODERM STRONG (Experimental): THIODERM STRONG injected into the upper arm (cohort 1)
  THIODERM STRONG injected into nasolabial folds (cohort 2)
  Interventions: Device: THIODERM STRONG

INTERVENTIONS:
Device: THIODERM STRONG — Soft tissue filler containing crosslinked hyaluronic acid and Na-hyaluronate, supplemented with lidocaine hydrochloride as ancillary substance.

SUMMARY:
This is a prospective, open label, dose-escalating, multicenter clinical investigation to evaluate the safety and effectiveness of THIODERM STRONG in the correction of nasolabial folds.

The performance is assessed using the 5-point Nasolabial Folds Severity Rating Scale (NLF-SRS) at Week 12 compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential must have a negative urine pregnancy test at Screening/ Baseline visit and must agree to use an adequate method of contraception for the duration of the clinical investigation
* Signed informed consent
* Moderate to severe nasolabial folds (cohort 2)
* Healthy skin in the nasolabial area and free of diseases that could interfere in cutaneous aging evolution (cohort 2)
* Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of the clinical investigation

Exclusion Criteria:

* For females: pregnant and/ or lactating or planning to become pregnant during the investigation
* History of allergies or hypersensitivity to hyaluronic acid preparations, lidocaine or any amide-basede anesthetic
* Tendency to keloid formation and/ or hypertrophic scars
* Presence of infectious, inflammatory or proliferative cancerous or pre-cancerous lesions in the area to be treated
* Recurrent herpes simplex in the treatment area
* History or presence of any autoimmune or connective tissue disease, or current treatment with immunomodulating therapy
* Diabetes mellitus or uncontrolled systemic diseases
* History of bleeding disorder and/ or use of anticoagulant, antiplatelet or thrombolytic medication from ten days pre- to three days post-injection
* Any medical condition prohibiting the inclusion in the clinical investigation according to the judgment of the investigator
* Previous enrollment in this clinical investigation
* Current participation in another clinical investigation, or treatment with any investigational drug/ medical device within 30 days prior to clinical investigation enrollment, or five half-lives of the investigational drug, whichever is longer
* Any dependency of the subject to the investigator or investigation site, or subjects who are employees or relatives of the investigator
* Subjects whose participation in clinical investigations is prohibited by the Austrian Medical Devices Act
* Facial plastic surgery, tissue augmentation with silicone, fat or another non-absorbable substance in the area of device application (cohort 2)
* Implantation of facial dermal fillers in the treatment area in the preceding 12 months (cohort 2)
* Skin of the nasolabial region affected by aesthetic treatments or planning to undergo such procedures during the clinical investigation (cohort 2)
* Facial lipolysis, including submental fat treatments within last month prior to enrollment or planned during the clinical investigation (cohort 2)
* Bariatric surgery within 12 months prior to enrollment or planned during the clinical investigation (cohort 2)
* Planned dental/ oral surgery or modification within two weeks prior to injection and to a minimum of four weeks post injection (cohort 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Frequency, severity, seriousness and causal relationship of AEs | Up to 4 weeks
Cohort 1: Local tolerability assessment based on presence and intensity of erythema, swelling and skin hardening | Up to 4 weeks
  5-grade scale ranging from 0 (absent), over 1 (minimal), 2 (mild), 3 (moderate), to 4 (severe)
Cohort 2: Improvement of at least 1 point on the Nasolabial Folds Severity Rating Scale (NLF-SRS) based on investigator's live assessment | Week 12 compared to baseline
  Scale from 0 (=none/ minimal) to 4 (= extreme)

SECONDARY OUTCOMES:
Cohort 2: Response rate based on investigator's assessment of Nasolabial Folds Severity Rating Scale (NLF-SRS) | Week 4, 24, 36 and 52 compared to baseline
  Scale from 0 (=none/ minimal) to 4 (= extreme)
Cohort 2: Gloabl aesthetic improvement scale (GAIS) determined by the investigator | Week 4, 12, 24, 36 and 52 compared to baseline
  global aesthetic improvement rated as 'very much improved', 'much improved', 'improved', 'no change' or 'worse'
Cohort 2: Gloabl aesthetic improvement scale (GAIS) determined by the subject | Week 4, 12, 24, 36 and 52 compared to baseline
  global aesthetic improvement rated as 'very much improved', 'much improved', 'improved', 'no change' or 'worse'
Cohort 2: Subject satisfaction based on Face-Q questionnaire "Satisfaction with Outcome" Scale | Week 4, 12, 24, 36 and 52 compared to baseline
Cohort 2: Response rate based on blinded photographic reviewer's assessment of Nasolabial Folds Severity Rating Scale (NLF-SRS) | Week 4, 12, 24, 36 and 52 compared to baseline
  Scale from 0 (=none/ minimal) to 4 (= extreme)
Cohort 2: Response rate based on investigator's assessment of Nasolabial Folds Severity Rating Scale (NLF-SRS) | Week 4, 12, 24, 36 and 52 compared to baseline
  Scale from 0 (=none/ minimal) to 4 (= extreme)
Cohort 2: Mean pain intensity score using the Numeric Pain Rating Scale (NPRS) | Immediately after administration and 15 minutes after treatment
  11-point scale ranging from 0 (= no pain) to 10 (=worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Medizinsche Universität Graz-Klinikum für Dermatologie und Venerologie, Graz
  - Yuvell, Vienna